CLINICAL TRIAL: NCT00821041
Title: Evaluation of an Internet-based Treatment for Chronic Insomnia
Brief Title: Internet-based Treatment for Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Nora Vincent, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2004:112; HSCF 176
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Insomnia; Insomnia Disorder
Keywords: insomnia; online systems
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list control (No Intervention)
- CBT (Experimental): A 6 weeks online course. Each week participants log on to view videos and read information that focus on a variety of intervention techniques. These include relaxation training, cognitive therapy, sleep restriction, stimulus control, sleep hygiene, psychoeducation, hypnotic tapering and mindfulness training. Participants also monitor their sleep using an online sleep diary and respond to questions regarding their adherence to the program.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 6 weeks of relaxation training, cognitive therapy, sleep restriction, stimulus control, sleep hygiene, psychoeducation, hypnotic tapering and mindfulness training
  Other Names: CBT
  Arms: CBT

SUMMARY:
Study Objectives. Despite effective cognitive behavioral treatments for chronic insomnia, such treatments are underutilized. This study evaluates the impact of a 6-week, online treatment for insomnia.

Design This is a randomized controlled trial with online treatment and waiting list control conditions.

Participants

Participants are adults in Manitoba Canada with chronic insomnia.

Setting

Participants receive online treatment from their homes. Intervention. Online treatment consists of psychoeducation, sleep hygiene and stimulus control instruction, sleep restriction treatment, mindfulness training, relaxation training, cognitive therapy, and help with medication tapering. Measurement and Results. The impact of online treatment on primary end points of sleep quality, insomnia severity, and daytime fatigue will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Access to high speed internet, insomnia duration > 6 months and occurring at least 4 nights per week, sleep-onset latency > 30 minutes and/or time awake at night > 30 minutes, and/or early morning awakening > 30 minutes before desired time, at least one type of daytime impairment.

Exclusion Criteria:

* Shift work, acute suicidality, mania, schizophrenia, head injury, alcohol intake > 14 drinks/week for males, > 12 drinks per week for females, current or past behavioral treatment for insomnia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-09; Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norah Vincent, Ph.D., Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Vincent N, Walsh K, Lewycky S. Determinants of success for computerized cognitive behavior therapy: examination of an insomnia program. Behav Sleep Med. 2013;11(5):328-42. doi: 10.1080/15402002.2012.700662. Epub 2013 Jan 3. PMID 23286463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Waiting List Control | Cognitive Behavioral Therapy
Started | 59 | 59
Completed | 59 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Waiting List Control | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 59 | 59 | 118
Age Continuous [Mean (Standard Deviation); unit: Years] | 50.45 (13.26) | 48.56 (11.39) | 49.54 (12.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 20 | 19 | 39
Total Sleep Time [Mean (Full Range); unit: Hours] — Total sleep time is collected from patients self-report weekly sleep diaries. It is the length of time spent in bed minus sleep onset latency and time spent awake in bed.
  Hours | 5.54 [1.74 to 10.80] | 5.61 [1.73 to 10.35] | 5.58 [1.73 to 10.80]

OUTCOME MEASURES:

1. Primary Outcome: Sleep Quality
Description: Sleep Quality was assessed by taking the average of two items: "How well do you feel this morning?" And "How enjoyable was your sleep last night?" (0 = not at all, 4 = very).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: 0-4 scale of sleep quality
Arm/Group | Waiting List Control | Cognitive Behavioral Therapy
Number analyzed (Participants) | 59 | 59
0-4 scale of sleep quality | 1.77 (0.77) | 2.18 (0.87)

2. Secondary Outcome: Pre-Sleep Arousal
Description: Pre-sleep Arousal Scale (cognitive subscale). 8-item measure of cognitive hyperarousal associated with insomnia. The subscale score can range from 8 to 40, with higher scores indicating more hyperarousal.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: PSA Scale
Arm/Group | Waiting List Control | Cognitive Behavioral Therapy
Number analyzed (Participants) | 59 | 59
PSA Scale | 25.46 (7.53) | 22.42 (7.97)

3. Secondary Outcome: Beliefs and Attitudes About Sleep
Time Frame: 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Waiting List Control | Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes